CLINICAL TRIAL: NCT05681910
Title: Predictive Factors for Mode of Extraction of the Uterus in Total Laparoscopic Hysterectomy
Brief Title: Mode of Uterine Extraction in Total Laparoscopic Hysterectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Gennaro Scutiero, MD, Università degli Studi di Ferrara
Other Study IDs: 879/2022/Oss/AOUFe
Record Dates: First submitted 2023-01-03; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hysterectomy remains the most common major gynecological operation worldwide. It may be carried out by three different routes and its variations: vaginal, abdominal, and laparoscopic.

A large uterus will lead to several surgical difficulties during laparoscopic hysterectomy, such as limited operative field, restrictive instrument range of motion, and difficult removal of the specimen.

The aim of this study was to compare the clinical results of TLH for large uterus through transvaginal or uterine morcellation approaches after strict preoperative assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total laparoscopic hysterectomies for larger uteri

Exclusion Criteria:

* oncology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinical data of patients undergoing total laparoscopic hysterectomies for larger uteri with uterus size of 12 gestational weeks (g.w.) or greater between. Inclusion criteria were as follows: (1) patients with uterine myomas or endometrioma; (2) patients who have good physical conditions and have no reproduction requirement; (3) patients with uterine size ≥ 12 weeks of gestation; and (4) patients who receive no hormone therapy in the recent 3 months. Exclusion criteria were as follows: (1) patients who are contraindicated to laparoscopic surgery; (2) patients with uterus size >16 g.w.; (3) patients with cervical myoma; (4) patients with uterine myoma associated with ovarian lesions; (5) patients with suspicious malignant gynecological disease diagnosed by ultrasound or MRI; and (6) patients with cervical cancer diagnosed by Thinprip cytologic test (TCT) and malignant endometrial lesions diagnosed by diagnostic curettage
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative complications | During surgery
  mean operation time, uterus removal time, blood loss
Post operative complications | 30 days after surgery
  Pelvic hematoma, vaginal stump infection, lower limb venous thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Obstetrics and Gynecology, Department of Morphology, Surgery and Experimental Medicine, University of Ferrara, Ferrara, Italy, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No